CLINICAL TRIAL: NCT01064674
Title: Cardiovascular Diagnostic Before Renal Transplantation: a Prospective Study to Assess Cardiovascular Morbidity Before Renal Transplantation and to Improve Standard Diagnostic Procedures.
Brief Title: Cardiovascular Evaluation Before Renal Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: PD Dr. med. Barbara Suwelack, Internal Medicine D, University Hospital of Muenster
Other Study IDs: KVDiagnostikpratransplantation; HerzundNierenMünster (Registry Identifier: clinical trials registry.)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Kidney Disease; Coronary Artery Disease
Keywords: renal transplantation; cardiovascular morbidity; evaluation before renal transplantation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- before renal transplantation: Patients with CKD IV° to V° who are actually registering for a renal transplantation in our department.
  Interventions: Other: diagnostic procedure

INTERVENTIONS:
Other: diagnostic procedure — Cardiovascular diagnostic standard procedure before renal transplantation using stress echocardiography and stress myocardial scintigraphy.
  Other Names: diagnostic standard procedure

SUMMARY:
Due to rising importance of cardiovascular disease before and after renal transplantation we have changed our standard diagnostic procedure and perform stress echocardiography and myocardial scintigraphy. We would like to monitor these results and the outcome of our patients.

DETAILED DESCRIPTION:
Chronic kidney disease is a well-known risk factor for cardiovascular disease. Patients waiting for a renal transplantation usually undergo an extensive diagnostic procedure to avoid complications after transplantation such as neoplasia or inflammation. In the past years, cardiovascular complications before and after renal transplantation have gained more attention. We therefore have changed our standard diagnostic procedure before renal transplantation and perform stress echocardiography and myocardial scintigraphy. Thus we would like to evaluate our new standard diagnostic procedure and observe the results of these diagnostic procedures as well as their impact on clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* endstage renal disease
* preparing for renal transplantation

Exclusion Criteria:

* children (< 18 years)
* women who are pregnant or nursing
* patients who are also awaiting heart transplantation or have already a heart transplant
* severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with endstage renal disease which are awaiting their ergsitration to our transplantation programm since July 2009 until July 2010.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
cardiovascular morbidity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Suwelack, MD, Principal Investigator — University Hospital Muenster; Hermann Pavenstädt, MD, Study Chair — University Hospital Muenster; Holger Reinecke, MD, Study Chair — University Hospital Muenster; Otmar Schober, MD, PhD, Study Chair — University Hospital Muenster
Locations (1):
- Department of Internal Medicine D, University Hospital Muenster, Münster, Germany